CLINICAL TRIAL: NCT04254926
Title: " Revie ⊕" Impact of a Resource-based Life Review Intervention on Patients With Advanced Cancer in an Outpatient Oncology Center: a Waitlist Randomized Controlled Trial
Brief Title: Impact of a Resource-based Life Review Intervention on Advanced Cancer Patients
Acronym: Revie⊕
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Collaborators: Krebsforschung Schweiz, Bern, Switzerland (Other); University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Gora Da Rocha, Professor assistant, School of Health Sciences Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KFS-4390-02-2018
Record Dates: First submitted 2019-12-14; First posted 2020-02-05 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Advanced Cancer
Keywords: resource-based; self-esteem; life review intervention

STUDY DESIGN:
Intervention Model Description: A pragmatic, two-arm parallel-group, waitlist randomized controlled trial (WLRCT) is conducted in which participants are randomized into (i) intervention, or (ii) waitlist control groups. The intervention group (IG) receives the Revie ⊕ intervention early on and the control group (CG) the same intervention but later on (i.e., after eight weeks).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Revie ⊕ intervention early (Experimental): participants randomized into (i) the intervention group (IG) receive the Revie ⊕ intervention early on.
  Interventions: Behavioral: Revie ⊕
- Revie ⊕ intervention later (Experimental): The control group (CG) receives the same intervention Revie ⊕ but later on (i.e., after eight weeks).
  Interventions: Behavioral: Revie ⊕

INTERVENTIONS:
Behavioral: Revie ⊕ — Revie ⊕ is a positive approach centered on the resources and strengths of the patient, and it consists of an intervention that focuses on the individual's life review. Revie ⊕ allows specialist nurses to discuss life events with cancer patients, to identify the significant elements, and to explore how the diagnosis has changed their values and preferences. The intervention is geared toward working with the patient to discover their potential, to identify their strategies for coping with the events of their life, and to thereby accompany them in achieving a better understanding of themselves and what defines their identity. The intervention also allows their concerns surrounding death to be addressed, in addition to providing clarity in regard to the life projects. In the end, as a conclusion to the intervention, the patient is provided a booklet recounting the salient features of their life review along with photographs, quotes, or images.

SUMMARY:
The main objective of the present study is to evaluate the effects of the Revie ⊕ intervention on the self-esteem of patients diagnosed with an advanced cancer. A pragmatic, two-arm parallel-group, waitlist randomized controlled trial is conducted. The study takes place in the oncology department of the University Hospitals of Geneva at 3 outpatient units.

DETAILED DESCRIPTION:
The main objective of the present study is to evaluate the effects of the Revie ⊕ intervention on the self-esteem of patients diagnosed with an advanced cancer. The secondary objectives are to evaluate the effects of the Revie ⊕ intervention on spiritual well-being, personal development, life satisfaction, and the perception of the interaction with the nurses. A pragmatic, two-arm parallel-group, waitlist randomized controlled trial (WLRCT) is conducted in which participants are randomized into (i) intervention, or (ii) waitlist control groups. The intervention group (IG) receives the Revie ⊕ intervention early on and the control group (CG) the same intervention but later on (i.e., after eight weeks).This monocentric study takes place in the oncology department of the University Hospitals of Geneva (HUG) at two outpatient units (planned n=102; 51 per group).

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years with and advanced cancer,
* whose general health status is adequate for participation in the study based on a clinical assessment by the nurse / doctor; and
* who consent to participate in the study.

Exclusion Criteria:

* documented cognitive impairment that compromises capacity for discernment,
* command of French is insufficient for reading, writing, or conversing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-04-06 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Self-esteem | Baseline, change from Baseline at 2 months, change from Baseline at 4 months
  Self-esteem will be measured by the Rosenberg Self-Esteem Scale (RSE, 10 items) developed in 1965 (French version).
  Minimum value = 1 Maximum value = 4. A score above 30 points corresponds to a high level of self-esteem, between 20 and 30 points indicates a moderate self-esteem, and a score of less than 20 points reflects a low self-esteem.

SECONDARY OUTCOMES:
Spiritual well-being | Baseline, change from Baseline at 2 months, change from Baseline at 4 months
  Spiritual well-being will be measured by the Functional Assessment of Chronic Illness Therapy-spiritual well-being (FACIT-Sp).
  Minimum value = 0 Maximum value = 4. The higher the score, the better the spiritual well-being.
Personal development | Baseline, change from Baseline at 2 months, change from Baseline at 4 months
  Personal development will be measured by the Post-Traumatic Growth Inventory (PTGI) instrument developed by Tedeschi and Calhoun in 1996 Minimum value = 1 Maximum value = 6. A high score means a high level of development.
Satisfaction with life | Baseline, change from Baseline at 2 months, change from Baseline at 4 months
  Satisfaction with life will be measured with the Satisfaction With Life Scale (SWLS) instrument developed by Pavot and Diener in 1985.
  Minimum value = 1 Maximum value = 7. A high score means a high level of satisfaction with life.
The patient's perception of their interaction with the nurse | Baseline, change from Baseline at 2 months, change from Baseline at 4 months
  The Nurse-Patient-Interaction Scale (NPIS) questionnaire developed by Haugan in 2012 will be used to evaluate the patient's perception of their interaction with the nurse Minimum value = 1 Maximum value = 10. A high score means a great appreciation of interaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Pautex, Professor, Principal Investigator — University Hospital, Geneva
Locations (2):
- Switzerland (2):
  - Hopitaux Universitaires de Genève, Geneva
  - Haute école de santé, Geneva

IPD SHARING:
Plan to Share IPD: No
this has to be specified later

REFERENCES:
- [Background] da Rocha Rodrigues MG, Pautex S, Zumstein-Shaha M. Revie plus sign in circle: An intervention promoting the dignity of individuals with advanced cancer: A feasibility study. Eur J Oncol Nurs. 2019 Apr;39:81-89. doi: 10.1016/j.ejon.2019.01.006. Epub 2019 Jan 30. PMID 30850142
- [Background] Da Rocha Rodrigues MG, Colin S, Shaha M, Pautex S. [The acceptability of the intervention Revie plus sign in circle : the nurses' perceptions and experiences]. Rech Soins Infirm. 2016 Dec;(127):55-70. doi: 10.3917/rsi.127.0055. French. PMID 28186482
- [Background] Da Rocha Rodrigues MG, Pautex S, Shaha M. Revie plus sign in circle: the influence of a life review intervention including a positive, patient-centered approach towards enhancing the personal dignity of patients with advanced cancer-a study protocol for a feasibility study using a mixed method investigation. Pilot Feasibility Stud. 2016 Oct 19;2:63. doi: 10.1186/s40814-016-0101-z. eCollection 2016. PMID 27965878
- [Derived] Da Rocha Rodrigues G, Warne DW, Scuderi L, Lilla D, Stanic J, Pautex S. Revie plus sign in circle: Impact of a resource-based life review intervention on patients with advanced cancer: A waitlist controlled trial. Eur J Oncol Nurs. 2024 Feb;68:102506. doi: 10.1016/j.ejon.2024.102506. Epub 2024 Jan 6. PMID 38301385